CLINICAL TRIAL: NCT03873922
Title: Dietary Intervention for Psychotic Disorders: a Pilot Intervention Study of Ketogenic Diet for Psychotic Symptoms - PsyDiet Pilot Study
Brief Title: Ketogenic Diet for Psychotic Disorders
Acronym: PsyDiet
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kuopio University Hospital (Other)
Collaborators: Deakin University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KUH5703458
Record Dates: First submitted 2018-08-28; First posted 2019-03-14 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Psychosis; Acute; Psychosis; Psychotic Disorders; Schizophrenia
Keywords: Ketogenic diet; Intervention; Ketosis; Feasibility; Psychosis; Psychotic symptoms; Schizophrenia; Dietary intervention
MeSH Terms: conditions — Psychotic Disorders; Schizophrenia; Ketosis

STUDY DESIGN:
Intervention Model Description: After baseline examinations, participants will be randomized to receive either ketogenic meals or conventional hospital meals during the study (maximum of six weeks). Otherwise treatment as usual.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Blinded research assistant will carry out the PANSS assessment and do the SCID-interviews. Care provider will order the meals for the participants, according to the randomization of the patients.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ketogenic diet intervention (Experimental): Ketogenic meals will be offered for the participants during the trial.
  Interventions: Other: Ketogenic diet intervention
- Control group (No Intervention): Conventional hospital meals as usual will be offered during the trial.

INTERVENTIONS:
Other: Ketogenic diet intervention — Ketogenic, really low carbohydrate containing (15-20 g/day), meals will be offered to the participants.
  Other Names: KD; Modified Ketogenic Diet
  Arms: Ketogenic diet intervention

SUMMARY:
Disturbances in glucose metabolism and glutamate neurotransmission feature in the pathophysiology of psychotic disorders. Ketogenic diet (KD) is a high-fat, low-carbohydrate diet that restricts glucose and forces metabolism of ketones, which serve as alternative energy substrates for the brain. KD is an established treatment for intractable epilepsy. However, we lack the randomized controlled trials (RCT) evidence regarding potential effects of KD on psychotic symptoms in humans.

This randomised, controlled pilot study aims to investigate:

1. feasibility of a Modified Ketogenic Diet (MKD) intervention protocol in psychotic inpatients,
2. potential impact of MKD intervention on psychotic symptoms, depressive and anxiety symptoms, and functioning in patients with psychotic symptoms / psychotic disorder.

A 6-week randomised KD pilot study will be carried out in psychotic inpatients (aimed n=40) at Niuvanniemi Hospital and Kuopio University Hospital, Finland. In the KD group, carbohydrate consumption is limited to 15-20 g/day to activate ketosis. The control group will have their ordinary hospital meals. A number of different assessment will be carried out at time points 0, 1 week, 3 weeks and 6 weeks.

DETAILED DESCRIPTION:
Disturbances in glucose metabolism and glutamate neurotransmission feature in the pathophysiology of psychotic disorders. Ketogenic diet (KD) is a high-fat, low-carbohydrate diet that restricts glucose and forces metabolism of ketones, which serve as alternative energy substrates for the brain. KD is an established treatment for intractable epilepsy. However, we lack the RCT evidence regarding potential effects of KD on psychotic symptoms in humans.

This randomised, controlled pilot study aims to investigate:

1. feasibility of a Modified Ketogenic Diet (MKD) intervention protocol in psychotic inpatients,
2. potential impact of MKD intervention on psychotic symptoms, depressive and anxiety symptoms, and functioning in patients with psychotic symptoms / psychotic disorder.

A 6-week randomised KD pilot study will be carried out in psychotic inpatients (aimed n=40) at Niuvanniemi Hospital and Kuopio University Hospital, Finland. In the KD group, carbohydrate consumption is limited to 15-20 g/day to activate ketosis. The control group will have their ordinary hospital meals. The Structured Clinical Interview for DSM Axis I disorders (SCID-I), and the Positive and Negative Syndrome Scale (PANSS) will assess current psychotic disorders and psychotic symptoms, respectively. Blood glucose, lipid, and ketone body levels, and weight will be measured. Background variables (socioeconomic factors, comorbidities, obtained treatments including medications, and health behaviours including diet) will be documented.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years old patient with psychotic symptoms / diagnosed psychotic disorder (ICD-10 diagnoses F20-F29)

Exclusion Criteria:

* BMI <18.5
* Diabetes mellitus (with or without insulin treatment)
* Inability to provide informed consent or to participate due to acute medical conditions, such as severe and acute psychotic symptoms or acute suicidality
* Impairments in vision, audition or immobility
* Pregnancy
* Diagnosed current eating disorder
* Diagnosed Inflammatory Bowel Disease (IBD)
* Severe alcohol or substance abuse
* Decompensated cardial insufficiency
* Infrequent/rare metabolic disorders, such as porphyria, disturbances in fatty acid oxidation or deficiency of CTT1, CPTII, carnitine or pyruvate carboxylase
* changes have occurred in psychotropic medications during the last 4 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-03-15 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
The change in Positive and Negative Syndrome Scale (PANSS) total score from baseline to 6 weeks. | The change from baseline to the end of the intervention (6 weeks) OR if discharged earlier, from baseline to the latest study assessment time point (1 or 3 weeks)
  Change in positive and negative psychotic symptoms, assessed at time points baseline, 1, 3 and 6 weeks. The participants are rated from 1 to 7 on 30 different symptoms based on the interview. PANSS Total score minimum is 30, maximum is 210. As 1 rather than 0 is given as the lowest score for each item, a participant can not score lower than 30 for the total PANSS score. Scores are given separately for the positive items, negative items, and general psychopathology scales which altogether (summarized) create a total PANSS score. Higher values represent a worse outcome.
Feasibility 1, defined by modified ketogenic diet related experiences, challenges and potential adverse effects during the intervention | Potential adverse effects during the entire trial will be evaluated (from baseline to 1, 3 and 6 weeks), as observed adverse effects may vary between study time points and status of ketosis
  Feasibility will be assessed by modified ketogenic diet related experiences, challenges and potential adverse effects by a Questionnaire of potential side effects and acceptance of MKD during the trial.
Feasibility 2, defined by percentage of study participants who discontinue diet and percentage of participants reaching ketosis (measured by blood ketone body levels) | Percentage of participants reaching ketosis and staying in ketosis in the MKD group will be calculated at each time point (weeks 1, 3 and 6)
  We will screen blood ketone body levels daily (MKD participants) or weekly (control participants). If participants in the MKD arm are not able to adhere to MKD, they will not reach ketosis or will not stay in ketosis. Feasibility will be defined by percentage of study participants reaching ketosis in the MKD group. In addition, drop-out rate of participants in each study arm will be calculated.

SECONDARY OUTCOMES:
The change in Beck Depression Inventory (BDI) score from baseline to 6 weeks. | Change in BDI score from baseline to 6 weeks OR if discharged earlier, from baseline to the latest study assessment time point (3 weeks)
  Change in depressive symptoms assessed by Beck Depression Inventory scores. BDI is a series of questions developed to measure the intensity, severity, and depth of depression in patients with psychiatric diagnoses. It is composed of 21 questions, each designed to assess a specific symptom. each with four possible responses. Each response is assigned a score ranging from zero to three, indicating the severity of the symptom. Score range is 0-63. Higher values represent a worse outcome.
The change in Beck Anxiety Inventory (BAI) score from baseline to 6 weeks | Change in BAI score from baseline to 6 weeks OR if discharged earlier, from baseline to the latest study assessment time point (3 weeks)
  Change in anxiety symptoms assessed by BAI scores. BAI evaluates both physiological and cognitive symptoms of anxiety and item overlap with other self report depression inventories is minimised. The BAI consists of 21 items; each item is descriptive of a symptom of anxiety and is rated on a scale of 0 to 3. Thus, the score range is from 0 to 63. Higher values represent a worse outcome.
The change in Structured Clinical Interview for DSM Axis I disorders (SCID-I) diagnosis from baseline to 6 weeks | Change in SCID-I diagnosis from baseline to 6 weeks
  The Structured Clinical Interview for DSM Axis I disorders assessing psychotic symptoms (SCID-I) is a validated semi-structured clinical interview (the gold standard tool for psychiatric assessment in a research setting). SCID-I will be used to assess for past and current psychotic disorders at the beginning and at the 6 week of intervention.
The change in the Global Assessment of Functioning score from baseline to 6 weeks. | Change in GAF score from baseline to 6 weeks OR if discharged earlier, from baseline to the latest study assessment time point (1 or 3 weeks)
  Change in The Global Assessment of Functioning (GAF). GAF interview will be conducted at each study time point (baseline, 1, 3 and 6 weeks). GAF scale is used to rate how serious a mental illness may be. It measures how much a person's symptoms affect his or her day-to-day life on a scale of 0 to 100. Higher values represent a worse outcome.

OTHER OUTCOMES:
Change in Blood lipid levels | Change in blood lipids between baseline and 6 weeks
  Change in measurements of blood lipids (fP-Kol, fP-KOL-LDL, fP-KOL-HDL, fP-Trigly)
Change in Fasting glucose levels | Change in blood lipids between baseline and 6 weeks
  Change in measurement of fasting glucose
Change in weight/body mass index (BMI) from baseline to 6 weeks | Change in weight/BMI from baseline to 6 weeks OR if discharged earlier, from baseline to the latest study assessment time point (1 or 3 weeks)
  Change in measured weight/BMI
Change in blood pressure (diastolic and systolic) from baseline to 6 weeks. | Change in blood pressure from baseline to 6 weeks OR if discharged earlier, from baseline to the latest study assessment time point (3 weeks)
  Change in blood pressure (diastolic and systolic)

CONTACTS AND LOCATIONS:
Overall Officials: Anu Ruusunen, PhD, Principal Investigator — Kuopio University Hospital
Locations (1):
- Kuopio University Hospital, Department of Psychiatry, Kuopio, Finland

IPD SHARING:
Plan to Share IPD: Undecided
Will be decided shortly.